CLINICAL TRIAL: NCT06538402
Title: Ileal Reservoir Length and Functional Outcome in Ileal Pouch-anal Anastomosis
Brief Title: Ten Versus Fifteen Centimeter Pouch in IPAA Surgery
Acronym: TESTIMONY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OP_2227
Record Dates: First submitted 2024-08-01; First posted 2024-08-05 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Ulcerative Colitis; Familial Adenomatous Polyposis
Keywords: ileal pouch-anal anastomosis; ulcerative colitis; familial adenomatous polyposis; randomized controlled trial; pouch function; quality of life; complications
MeSH Terms: conditions — Colitis, Ulcerative; Adenomatous Polyposis Coli

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 cm (Experimental): Ileal reservoir length of 10 cm
  Interventions: Procedure: 10 cm pouch
- 15 cm (Active Comparator): Ileal reservoir length of 15 cm
  Interventions: Procedure: 15 cm pouch

INTERVENTIONS:
Procedure: 10 cm pouch — A 10 cm pouch will be constructed
  Arms: 10 cm
Procedure: 15 cm pouch — A 15 cm pouch will be constructed
  Arms: 15 cm

SUMMARY:
The aim of this randomized controlled trial is to compare outcome after construction of an ileal (J-shaped) reservoir of 10 versus 15 centimeters in primary ileal pouch-anal anastomosis surgery.

DETAILED DESCRIPTION:
The primary aim of this randomized controlled trial is to compare functional outcome in terms of bowel function correlated with quality of life for patients who undergo primary ileal pouch-anal anastomosis surgery with an ileal (J-shaped) reservoir length of either 10 cm or 15 cm.

Secondary aims include health-related quality of life measures and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing ileal pouch-anal anastomosis (IPAA) for ulcerative colitis or familial adenomatous polyposis (FAP) (implying a normal sphincter function as judged by history and clinical examination)
* Signed informed consent
* Able to perform both a small (10 cm) and medium-size (15 cm) pouch with adequate reach and no tension as determined subjectively by the surgeon intraoperatively

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2028-07-03 (Estimated); Study Completion 2038-07-03 (Estimated)

PRIMARY OUTCOMES:
Pouch dysfunction score | 1, 3, 5 and 10 years after surgery
  Ranges from 0 to 7.5, where a low score indicates good bowel function will little to no impact on quality of life

SECONDARY OUTCOMES:
Short Inflammatory Bowel Disease Questionnaire | 1, 3, 5 and 10 years after surgery
  Consists of 10 questions with a total score range from 10 (poor health-related quality of life) to 70 (good health-related quality of life)
Short-form (SF)-36 | 1, 3, 5 and 10 years after surgery
  Consists of questions relating to 8 domains of life with a total score ranging from 0-100, with lower numbers indicating worse health status
Postoperative complications using the Comprehensive Complication Index (CCI) | 90 days after surgery
  The CCI is a continuous scale, where each postoperative complication as defined by Clavien-Dindo is assigned a weigth based on its severity. A total summarized score taking all complications into account is thus generated.
Pouch failure | 1, 3, 5 and 10 years after surgery
  Hazard ratio of pouch failure defined as an intended permanent ileostomy with or without pouch excision

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Hvidovre Hospital, Hvidovre